CLINICAL TRIAL: NCT04377256
Title: Hyaluronic Acid Effect on Xenogenic Bone Substitutes Healing During Ridge Preservations: A Radiological and Histomorphometric Study
Brief Title: Hyaluronic Acid Effect on Xenogenic Bone Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: USJ-2019-267
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Bone Resorption; Tooth Loss
Keywords: tooth extraction; ridge preservation; hyaluronic acid; dental implant
MeSH Terms: conditions — Bone Resorption; Tooth Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiological assessement (Experimental): Two CBCTs were recorded and compared, one at the baseline and the other at 4 months post-op. The bone resorption was quantified and analyzed using ITK-SNAP software
  Interventions: Procedure: Ridge preservation: Tooth extration and immediat bone grafting in the socket
- Histomorphometric analysis (Experimental): During implant placement (4 months after the bone grafting), a bone biopsy is collected and stained with several colorants to analyze the biological bone healing
  Interventions: Procedure: Ridge preservation: Tooth extration and immediat bone grafting in the socket

INTERVENTIONS:
Procedure: Ridge preservation: Tooth extration and immediat bone grafting in the socket — Following the tooth extraction, the socket is filled with a mixture of xenogenic bone and hyaluronic acid and sealed with an epithelio-connective arrested from the maxillary palate

SUMMARY:
The aim of this study is to test the hyaluronic acid hydrogel impact on the healing acceleration of xenogenic bone substitutes used in ridge preservation.

Following tooth extraction, bone particles are mixed with the hyaluronic acid gel and grafted in the tooth socket. at the implant placement phase, a cone beam computer assisted tomography file is recorded in order to compare it with the baseline and a biopsy to evaluate the histological consequences.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of tooth extraction and willing to receive dental implants in the extraction site
* Presence of two mono radicular teeth in need of extraction

Exclusion Criteria:

* Patients with systemic diseases
* Patients under 8 years and above 60 years.
* Presence of endodontic or periodontal lesion in the extraction sites

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Radiological assessement of the boe resorption | 4 months
  the baseline if the CBCT is compared to the 4 months post-op to assess the bone resorption
Histomorphometric analysis | 4 months
  During implant placement, a bone biopsy is harvested and stained with different colorants to assess microscopically the biological healing

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Younes, Phd, Study Director — Head of oral surgery department, facuty of dentistry ,Universite SainT Joseph-Beyrouth; Bachar A Husseini, DDS, Principal Investigator — Department of oral surgery, facuty of dentistry ,Universite SainT Joseph-Beyrouth
Locations (2):
- Lebanon (2):
  - Saint-Joseph university, Beirut, Lebanon
  - Universte Saint Joseph-Beyrouth, Beirut

IPD SHARING:
Plan to Share IPD: No